CLINICAL TRIAL: NCT04866823
Title: Meals for Moms: A Postpartum Medically-Tailored Meal Program to Promote Weight Loss and Blood Glucose Control Among Women With Hyperglycemia in Pregnancy
Brief Title: Meals for Moms: Medically-Tailored Meals for Women Who Had Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: North Carolina Diabetes Research Center (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00072715; 40010554 (Other: National Institute of Diabetes and Digestive and Kidney Diseases)
Record Dates: First submitted 2021-04-26; First posted 2021-04-30 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2023-02

CONDITIONS: Diabetes, Gestational; Gestational Weight Gain; Postpartum Weight Retention
Keywords: Lifestyle Intervention; Weight-Loss; Self-Care
MeSH Terms: conditions — Diabetes, Gestational; Gestational Weight Gain; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medically Tailored Meals (Experimental): A series of medically tailored meals appropriate for women with gestational diabetes will be developed in partnership with chefs from a local community kitchen and catering company. Meals will create a slight caloric deficit in order to promote gradual weight loss, but with sufficient energy intake and macronutrient balance to allow breastfeeding. These meals will be roughly 40% carbohydrate, 30% protein, and 30% fat in composition. Study Team will plan up to 20 unique lunch and dinner meals for the series. Each meal will be prepared to be between 450-600 kcal and to contain 6 ounces of protein, 4 ounces of vegetable and I cup of whole grain (at a minimum). Participants will receive detailed recipe cards and nutrition information with each meal. In addition to receiving the medically tailored meals, participants will be advised to supplement their own breakfast +/- snacks to reach a total daily calorie goal determined by starting BMI category.
  Interventions: Behavioral: Medically Tailored Meals
- Usual Care Comparison Group (No Intervention): Participants in this group will receive written materials on self-care, nutrition, and physical activity in the postpartum period and community resources for healthy living.

INTERVENTIONS:
Behavioral: Medically Tailored Meals — Participants will receive weekly meals (20 per week) prepared by a local community kitchen and catering group. Each week, 10 dinners and 10 lunches will be delivered to the participant's home with instructions for storage, re-heating, recipes, and nutritional information.
  Arms: Medically Tailored Meals

SUMMARY:
The purpose of this research study is to test whether delivery of medically tailored meals (meals designed specifically to be healthy) can be used to help reduce high blood sugar after delivery of a baby. Participants will be recruited and consented during the third trimester of pregnancy but will begin study activities after delivery. Participants will complete a series of questionnaires on demographics, health history, home environment, overall and financial stress, plans for weight loss and infant feeding, and food insecurity. Participants will also be asked to wear continuous glucose monitors for two separate 14-day periods (within 2 weeks of delivery and at 3 months). All participants will receive weekly emails with educational videos and 3 virtual visits with a member of the study team and will also be randomly assigned to an intervention or comparison group. In the intervention, participants will receive weekly meal deliveries of 10 pre-prepared meals from Providence Community Kitchen (local company in Winston-Salem, NC) that are calorically restricted and appropriate for post-partum women with a history of gestational diabetes and who may be breast-feeding. Women in the control condition will receive written resources on self-care, nutrition, and physical activity appropriate for post-partum women who had gestational diabetes.

DETAILED DESCRIPTION:
Pregnancy and delivery can function as a "stress test" for future development of cardiovascular disease and metabolic disorders, with gestational diabetes and excessive weight gain during pregnancy leading to worse outcomes later in a mother's life. The prevalence of both conditions continues to increase with the obesity epidemic, highlighting the urgent need for successful interventions to reverse maternal weight gain and promote normal blood sugars. The early postpartum period provides a critical opportunity to address diet behaviors that are related to both weight and diabetes. Postpartum medically-tailored meal delivery is a novel approach that may allow for improved blood sugar control and weight loss in a traditionally hard-to-engage patient population. There is currently no available data on the cost, feasibility, or effectiveness of providing medically-tailored meals to postpartum women. This is a pilot study of medically-tailored meals for new mothers whose pregnancies were complicated by gestational diabetes, and whose total gestational weight gain exceeded recommendations. Study will enroll 30 women with gestational diabetes and excessive gestational weight gain late in the third trimester of a singleton pregnancy. Data collection and intervention activities will begin after delivery. All participants will wear a continuous glucose monitor for baseline (first 2 weeks after delivery) and at follow up (after 3 months). Participants will also completed self-administered questionnaires, receive weekly informational videos by email, and have 3 monthly in-person check-ins with a member of the study team. Twenty participants will be randomly assigned to a medically-tailored meals intervention and 10 to a usual-care comparison group. A local community-based program will prepare and deliver 10 medically-tailored meals per week to intervention participants for their first 3 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Demographics: Women 18 years of age and older who reside in Forsyth County, NC
* Pregnancy: Currently 24 or more weeks into a singleton pregnancy
* Clinical evidence of gestational diabetes mellitus (GDM) defined as either 3-hour oral glucose tolerance test (OGTT) results obtained in the second trimester of pregnancy that show at least 2 abnormal values or a diagnosis of "gestational diabetes" included on the Problem List in medical record during current pregnancy, regardless of OGTT values
* Excessive gestational weight gain: Most recent weight exceeds predicted weight gain for current weeks gestational age defined as pre-pregnancy Body mass index (BMI) of 30 kg/m2 or more and weight at most recent clinical visit 20+ pounds over pre-pregnancy weight or pre-pregnancy BMI of 25-29.9 kg/m2 and weight at most recent clinical visit 25+ pounds over pre-pregnancy weight
* English Proficiency: Able to read/understand English at or above a level sufficient to comprehend recruitment, informed consent, and intervention materials.
* Access to a smart phone/tablet/computer capable of connecting to video calls or teleconferencing software.
* Willingness to Accept Randomization: Prospective participants must be willing to accept randomization to either the medically tailored meal intervention or the comparison intervention condition.

Exclusion Criteria:

* Clinical history of diabetes (type 1 or 2) pre-pregnancy
* Non-singleton pregnancy
* Other chronic diseases or medical conditions that would increase risk or make participation otherwise unsafe, including special dietary needs. A clinician investigator will review the medical record for all potential participants to determine if any such conditions exist.
* Known food allergies of sensitivities. Potential participants who report special dietary requirements including vegetarians, vegans, those who follow kosher or other specialized diets will be excluded due to the small nature of this pilot study.
* History of allergic skin reaction to adhesive tape
* Unable or unwilling to wear a continuous glucose monitor (CGM) device
* Is scheduled for an MRI during the study weeks, making use of the CGM device unsafe
* Other: Conditions/criteria likely to interfere with participation and acceptance of randomized assignment, including the following: inability/unwillingness to give informed consent, major psychiatric or cognitive problems (schizophrenia, dementia, self-reported substance or alcohol abuse), participation in another research study that would interfere with Meals for Moms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants are required to be biological Females
Enrollment: 12 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morgana Mongraw-Chaffin, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to recruitment limitations, we did not include a comparison group.
Period: Overall Study
Arm/Group | Medically Tailored Meals | Usual Care Comparison Group
Started | 12 | 0 (Due to recruitment limitations, we did not include a comparison group.)
Completed | 9 | 0
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Due to recruitment limitations, we did not inlcude a comparison group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Medically Tailored Meals | Usual Care Comparison Group | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 12 |  | 12
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (5) |  | 35 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 |  | 12
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 |  | 6
  Not Hispanic or Latino | 6 |  | 6
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 2 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 5 |  | 5
  White | 3 |  | 3
  More than one race | 2 |  | 2
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Meals Successfully Ordered and Delivered
Description: Determine the percent of meals successfully ordered & delivered in the intervention group
Time Frame: 3 months
Population: No comparison group was included due to limited recruitment numbers.
Measure: Count of Units; unit: meals
Units Other Than Participants: meals
Arm/Group | Medically Tailored Meals | Usual Care Comparison Group
Number analyzed (Participants) | 12 | 0
Number analyzed (meals) | 2880 | 0
meals | 2880 |

2. Primary Outcome: Number of Dollars Cost
Description: Determine the total cost across all participants for the medically tailored meal program per participant assuming 20 meals per week provided to each participant for 12 weeks.
Time Frame: 3 months
Population: No comparison group was included.
Measure: Number; unit: Number of dollars cost
Arm/Group | Medically Tailored Meals | Usual Care Comparison Group
Number analyzed (Participants) | 12 | 0
Number of dollars cost | 1800.0 |

3. Primary Outcome: Days of Continuous Glucose Monitoring in Postpartum Mothers
Description: Tracking the number of days the continuous glucose monitors were worn (of 14 total possible) at baseline.
Time Frame: 14 day period assessed at baseline
Population: No comparison group was included.
Measure: Mean (Full Range); unit: Number of Days
Arm/Group | Medically Tailored Meals | Usual Care Comparison Group
Number analyzed (Participants) | 12 | 0
Number of Days | 13 [6 to 14] |

4. Primary Outcome: Days of Continuous Glucose Monitoring in Postpartum Mothers
Description: Tracking the number of days the continuous glucose monitors were worn (of 14 total possible) at 3 months.
Time Frame: 3 months
Population: No comparison group was included due to limited recruitment numbers.
Measure: Mean (Full Range); unit: days
Arm/Group | Medically Tailored Meals | Usual Care Comparison Group
Number analyzed (Participants) | 7 | 0
days | 11.43 [1 to 14] |

ADVERSE EVENTS:
Time Frame: 3 months
Description: No comparison group was included. All participants received the medically tailored meals.
Arm/Group | Medically Tailored Meals | Usual Care Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/0
Other Adverse Events (participants affected / at risk) | 0/12 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT04866823/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT04866823/ICF_000.pdf